CLINICAL TRIAL: NCT02277236
Title: Creating a Model of Proactive Geriatric Care Within VISN 5: Screening for Age-Related Skeletal Muscle Dysfunction at the Washington DC VA Medical Center
Brief Title: Screening for Age-Related Skeletal Muscle Dysfunction
Acronym: ARMS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harris-Love, Principal Investigator, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: MIRB01671
Record Dates: First submitted 2014-10-18; First posted 2014-10-28 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Sarcopenia
Keywords: sarcopenia; aging; insulin resistance; screening
MeSH Terms: conditions — Sarcopenia; Insulin Resistance | interventions — X-Rays; Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for determination of lipid profiles, fasting insulin and glucose levels, the oral glucose tolerance test, and selected cytokines (IL-6 and TNF-α).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Younger Veterans: Male Veterans, 45-64.9 years of age. (Exposures include DXA scanning and CT imaging.)
  Interventions: Radiation: DXA scanning; Radiation: CT imaging
- Young-Old Veterans: Male Veterans, 65-84.9 years of age. (Exposures include DXA scanning and CT imaging.)
  Interventions: Radiation: DXA scanning; Radiation: CT imaging

INTERVENTIONS:
Radiation: DXA scanning — Exposure: Participants will undergo DXA scanning in the supine position per manufacturer guidelines to estimate absolute and percentage of total lean body mass (LBM) and body fat (BF).
  Other Names: Radiograph, x-rays
Radiation: CT imaging — Exposure: Estimates of intramuscular adipose tissue (IMAT) will be obtained with CT imaging. This measure will be restricted to a single leg (dominant side) in the mid-femur region, using a single 10mm axial image slice (120 kVp, 200 to 250 mA).
  Other Names: CAT scan

SUMMARY:
This pilot study will aid the development of a sonographic screening method used to obtain proxy measures of LBM and estimates of muscle composition that relate to Intramuscular adipose tissue (IMAT), lipid metabolism, and insulin resistance. Typically, age-related muscle loss is not assessed in older adults until they began to show signs of trouble managing their own lives independently. In addition to the loss of independence that is typically seen with diminished muscle mass and function (sarcopenia), age-related changes in lean body mass can have negative effects on insulin sensitivity. The investigators central hypothesis is that the muscle characteristics derived from ultrasound (US) will be significantly associated with estimates of dual energy X-ray absorptiometry (DXA) LBM, CT scan measures of IMAT, estimates of insulin homeostasis, and serum levels of inflammatory cytokines.

DETAILED DESCRIPTION:
The primary goals of this project are to: 1) develop and validate a rapid, portable, cost-effective, screening method for sarcopenia using diagnostic ultrasound (US), and 2) determine if the US screening method provides viable estimates of intramuscular adipose tissue (IMAT) since muscle tissue age-related changes in muscle composition are associated with low muscle torque and metabolic dysfunction. The proposed US screening method may be used as a proxy measure of LBM and provide estimates of skeletal muscle composition that relate to IMAT, lipid metabolism, insulin homeostasis and inflammation - important factors that may impact impaired mobility and metabolic dysfunction in older African American Veterans.

Aim 1:

Determine the association between a proxy measure of LBM obtained via portable, diagnostic, musculoskeletal US and LBM as determined by dual energy X-ray absorptiometry (DXA).

The working hypothesis is that a 6-muscle model of LBM derived from US and DXA LBM values will exhibit a significant positive association and attain a coefficient of determination > .80.

Aim 2:

Determine the association between US echointensity features and IMAT as determined by CT scan.

US echointensity values will be acquired from the rectus femoris and analyzed to determine the association with IMAT. The working hypothesis is that higher echointensity values measured with grayscale analysis will be negatively associated with the Hounsfield units obtained from the CT scan (p < .05).

Aim 3:

Examine the association between US echointensity values and biologic factors that impair insulin sensitivity.

Excessive IMAT and intra-myocellular triglyceride levels result in increased levels of biologic factors such as inflammatory cytokines (TNF-α and IL-6), which may affect insulin sensitivity. The investigators hypothesis is that proxy measures of IMAT via echointensity values will be positively associated with biomarkers of inflammation and insulin homeostasis.

ELIGIBILITY:
Inclusion Criteria: You are eligible to participate if:

1. You are registered to receive healthcare at the Washington DC VAMC through the Geriatrics Extended Care Service and/or Primary Care Service.
2. You are a male.
3. You are between the ages of 45 - 85 years.
4. Must be able to stand comfortably for 10 minutes and walk a short distance (use of assistive devices are acceptable).

   -

Exclusion Criteria: You are not eligible to participate if:

1. You have uncontrolled hypertension.
2. Body Mass Index (BMI) <18.5 or >32.5.
3. Musculoskeletal conditions that would stop you from performing the physical assessment test.
4. Muscle weakness due to neurological disease or injury (such as stroke or spinal cord injury).
5. Moderate to severe sepsis (blood infection) or edema (such as swelling of a limb).
6. Currently prescribed medications that affect glucose or insulin.
7. Uncontrolled cardiovascular disease.
8. Hospitalization over the last three months.
9. Diagnosis of diabetes.

   -

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veteran men (45-85 years of age; n = 30) consecutively recruited from outpatients at the DC VAMC and assigned to a "younger" or "young old" group (i.e., 45-64.9, and 65-84.9 years of age).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Sonographic Lean Body Mass | 1 day
  US estimates of aggregate regional LBM (muscle thickness, cm), will be assessed using B-mode diagnostic US with a 13-6 MHz linear array transducer for morphology measures at 6 axial and appendicular sites. The following sites will be assessed: the midpoint of the upper trapezius, upper pectoralis major, lateral deltoid, brachioradialis, rectus femoris, and tibialis anterior.

SECONDARY OUTCOMES:
Metabolic status | 1 day
  A blood sample (60 cc) will be obtained after an 8-hour overnight fast: glucose and insulin levels will be assessed before and during a standard (75 g) 2 hour oral glucose tolerance test. Other laboratory values such as a standard lipid profile and selected cytokines (IL-6), will also be measured.
DXA lean body mass | At time of assessment
  Participants will undergo dual energy X-ray absorptiometry (DXA) scanning in the supine position per manufacturer guidelines to estimate absolute and percentage of total LBM, and body fat percentage (BF%).
Intramuscular adipose tissue assessment | 1 day
  Estimates of intramuscular adipose tissue (IMAT) will be obtained with CT imaging. A single, unilateral 10mm axial image slice (120 kVp, 200 to 250 mA) of the thigh will be obtained at the midfemur region (corresponding to the ultrasound scanning site).
Strength assessment | 1 day
  Grip strength will be assessed bilaterally; isokinetic knee extension/flexion torques will be obtained bilaterally using the Biodex System 4. Peak concentric torque (at 60º/s and 180º/s) will be obtained in a randomized fashion with subject positioning and stabilization per the Biodex Operations Manual.
Functional assessment | 1 day
  A standardized timed sit-to-stand test will be conducted (5 repetitions); 6m walking speed (habitual and fast gait) will be recorded; the Physical Performance Test (PPT-7), a functional battery validated for use with older adults, will be used in this study to assess the activities of daily living of the participants.
Physical activity questionnaire | 1 day
  Participants will also complete the International Physical Activity Questionnaire (IPAQ) to obtain an estimate of their customary activity and formal exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, MPT, DSc, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Harris-Love MO, Adams B, Hernandez HJ, DiPietro L, Blackman MR. Disparities in the consequences of sarcopenia: implications for African American Veterans. Front Physiol. 2014 Jul 7;5:250. doi: 10.3389/fphys.2014.00250. eCollection 2014. No abstract available. PMID 25071595
- [Background] Harris-Love MO, Monfaredi R, Ismail C, Blackman MR, Cleary K. Quantitative ultrasound: measurement considerations for the assessment of muscular dystrophy and sarcopenia. Front Aging Neurosci. 2014 Jul 14;6:172. doi: 10.3389/fnagi.2014.00172. eCollection 2014. No abstract available. PMID 25071570
- [Derived] Gollie JM, Harris-Love MO, Patel SS, Shara NM, Blackman MR. Rate of Force Development Is Related to Maximal Force and Sit-to-Stand Performance in Men With Stages 3b and 4 Chronic Kidney Disease. Front Rehabil Sci. 2021 Sep 28;2:734705. doi: 10.3389/fresc.2021.734705. PMID 34708217